CLINICAL TRIAL: NCT07291076
Title: ROSETTA HCC-206: An Open-Label, Multi-Center, Randomized Phase 1/2 Study of Pumitamig Alone or In Combination With Ipilimumab in Participants With First-Line Advanced or Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: A Study to Evaluate the Safety and Tolerability of Pumitamig Alone or In Combination With Ipilimumab in Participants With First-Line Advanced or Unresectable Hepatocellular Carcinoma (HCC) (ROSETTA HCC-206)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA266-0006; 2025-523602-33 (Other: EU CT Number); U1111-1327-4912 (Other: UTN)
Record Dates: First submitted 2025-12-17; First posted 2025-12-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: First line HCC; Unresectable HCC; Ipilimumab; Pumitamig
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ipilimumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1A (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Cohort 1B (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Cohort 2A (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Cohort 2B (Experimental)
  Interventions: Drug: Pumitamig; Drug: Ipilimumab
- Cohort 2C (Other)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Cohort 2D (Experimental)
  Interventions: Drug: Pumitamig

INTERVENTIONS:
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545
  Arms: Cohort 1A; Cohort 1B; Cohort 2A; Cohort 2B; Cohort 2D
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Cohort 1A; Cohort 1B; Cohort 2A; Cohort 2B
Drug: Atezolizumab — Specified dose on specified days
  Arms: Cohort 2C
Drug: Bevacizumab — Specified dose on specified days
  Arms: Cohort 2C

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Pumitamig alone or in combination with Ipilimumab in participants with first-line advanced or unresectable Hepatocellular Carcinoma (HCC)

ELIGIBILITY:
Inclusion Criteria

* Participants must have a histologically confirmed diagnosis of locally advanced or unresectable Hepatocellular Carcinoma (HCC).
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must have no prior systemic therapy for advanced/ unresectable HCC.
* Participants must have measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Exclusion Criteria

* Participants must not have significant bleeding or coagulation disorders or other obvious bleeding risk evidence.
* Participants must not have an organ transplant or autoimmune disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-10-15 (Estimated); Study Completion 2031-10-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 25 weeks
  Phase 1
Number of participants with serious adverse events (SAEs) (as per Common Terminology Criteria for Adverse Events v5 (CTCAE v5)) | Up to approximately 25 weeks
  Phase 1
Number of participants with AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria | Up to day 21
  Phase 1
Number of participants with AEs leading to discontinuation | Up to approximately 25 weeks
  Phase 1
Number of participants with AEs leading to death | Up to approximately 25 weeks
  Phase 1
Objective response (OR) (confirmed complete response (CR) or partial response (PR)) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 per investigator assessment | Up to week 48
  Phase 2

SECONDARY OUTCOMES:
Number of participants with AEs | Up to approximately 25 weeks
  Phase 2
Number of participants with SAEs (as per CTCAE v5) | Up to approximately 25 weeks
  Phase 2
Number of participants with treatment-related adverse events (TRAEs) | Up to approximately 25 weeks
  Phase 2
Number of participants with AEs leading to discontinuation | Up to approximately 25 weeks
  Phase 2
Number of participants with AEs leading to death | Up to approximately 25 weeks
  Phase 2
End of infusion concentration of Pumitamig | Up to day 21
  Phase 2
End of trough concentration of Pumitamig | Up to day 21
  Phase 2
Trough concentration of Ipilimumab | Up to day 21
  Phase 2
Incidence of anti-drug antibodies against Pumitamig | Up to 5 years
  Phase 2
Incidence of anti-drug antibodies against Ipilimumab | Up to 5 years
  Phase 2
Progression-free survival (PFS) by RECIST v1.1 per investigator assessment | Up to 4 years
  Phase 2
Duration of response (DOR) (confirmed by PR or CR) by RECIST v1.1 per investigator assessment | Up to 4 years
  Phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (46):
- United States (8):
  - Local Institution - 0070, Los Angeles, California
  - Local Institution - 0107, Chicago, Illinois
  - Local Institution - 0103, Hackensack, New Jersey
  - Local Institution - 0100, Great Neck, New York
  - Local Institution - 0080, Portland, Oregon
  - Local Institution - 0022, Nashville, Tennessee
  - Local Institution - 0102, Nashville, Tennessee
  - Local Institution - 0083, Seattle, Washington
- Australia (4):
  - Local Institution - 0040, Birtinya, Queensland
  - Local Institution - 0024, Camperdown
  - Local Institution - 0096, Melbourne
  - Local Institution - 0033, Wentworthville
- Chile (2):
  - Local Institution - 0064, Santiago, Santiago Metropolitan
  - Local Institution - 0106, Santiago Region Metropolitana, Santiago Metropolitan
- China (3):
  - Local Institution - 0075, Guangzhou, Guangdong
  - Local Institution - 0086, Xi'an, Shaanxi
  - Local Institution - 0078, Shanghai, Shanghai Municipality
- France (5):
  - Local Institution - 0056, Pessac, Aquitaine
  - Local Institution - 0059, Rennes, Ille-et-Vilaine
  - Local Institution - 0004, Grenoble, Isère
  - Local Institution - 0018, Saint Priest En Jarez, Pays de la Loire Region
  - Local Institution - 0003, Bobigny
- Germany (3):
  - Local Institution - 0031, Cologne, North Rhine-Westphalia
  - Local Institution - 0028, Kiel, Schleswig-Holstein
  - Local Institution - 0030, Frankfurt
- Italy (4):
  - Local Institution - 0109, Pisa, Tuscany
  - Local Institution - 0088, Milan
  - Local Institution - 0016, Pisa
  - Local Institution - 0046, Rozzano (MI)
- Poland (3):
  - Local Institution - 0021, Wroclaw, Lower Silesian Voivodeship
  - Local Institution - 0105, Warsaw, Masovian Voivodeship
  - Local Institution - 0020, Gdansk
- Singapore (2):
  - Local Institution - 0009, Singapore
  - Local Institution - 0012, Singapore
- South Korea (3):
  - Local Institution - 0027, Seongnam-si, Gyeonggi-do
  - Local Institution - 0013, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0011, Seoul, Seoul-teukbyeolsi
- Spain (2):
  - Local Institution - 0014, Pamplona, Navarre
  - Local Institution - 0060, Madrid
- Taiwan (4):
  - Local Institution - 0032, Taichung
  - Local Institution - 0055, Tainan, Taiana
  - Local Institution - 0006, Taipei
  - Local Institution - 0007, Taipei
- United Kingdom (3):
  - Local Institution - 0073, London, London, City of
  - Local Institution - 0051, Glasgow, South Western Scotland
  - Local Institution - 0053, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07291076.html